CLINICAL TRIAL: NCT02498171
Title: Evaluation Of Efficacy And Safety Of Labour Analgesia By Intrathecal Morphine With Fentanyl Compared To Morphine With Bupivacaine In Mulago Hospital: A Double-blinded Randomized Control Trial
Brief Title: Labour Analgesia; Comparing a Combinations of Either Fentanyl or Bupivacaine With Intrathecal Morphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011/HD07/2061U
Record Dates: First submitted 2015-07-07; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Labor Pain
Keywords: Labour analgesia; Intrathecal morphine; Bupivacaine; Fentanyl
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl; Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal morphine with fentanyl (Experimental): Single shot of intrathecal morphine 100mcg mixed with 25mcg of fentanyl and filled up to make a 2ml solution. This would then be injected into the subarachnoid space through L2-3 or L3-4 following standard procedures.
  Interventions: Drug: Intrathecal morphine with fentanyl
- Intrathecal morphine with bupivacaine (Active Comparator): Single shot of intrathecal morphine 100mcg mixed with 2.5mg of spinal bupivacaine and filled up to make a 2ml solution.This would then be injected into the subarachnoid space through L2-3 or L3-4 following standard procedures.
  Interventions: Drug: Intrathecal morphine with bupivacaine

INTERVENTIONS:
Drug: Intrathecal morphine with fentanyl — Parturients in this arm underwent a single shot spinal following standard procedure. the drug mixture was then introduced into the subarachnoid space following free flow of csf. the parturient was the monitored fo labour progression using the standard partogram, vital signs and the visual analogue scale score for pain recorded every 5 min.
  The fetus was monitored with an ultrasonic aided fetal Doppler until delivery
  Other Names: Morphine Sulphate 10mg/ml, Ampoule 1ml,Martindale Hong Kong; Fentanyl Citrate 0.05mg/ml, Ampoule 2ml,Martindale Hong Kong
  Arms: Intrathecal morphine with fentanyl
Drug: Intrathecal morphine with bupivacaine — Parturients in this arm underwent a single shot spinal following standard procedure. the drug mixture was then introduced into the subarachnoid space following free flow of csf. the parturient was the monitored fo labour progression using the standard partogram, vital signs and the visual analogue scale score for pain recorded every 5 min.
  The fetus was monitored with an ultrasonic aided fetal Doppler until delivery
  Other Names: Morphine Sulphate 10mg/ml, Ampoule 1ml, Martindale Hong Kong; sesorcaine 0.5%, Ampoule 4ml, Astrazeneca
  Arms: Intrathecal morphine with bupivacaine

SUMMARY:
This study is aimed at evaluating single short spinal technique as a form of labour analgesia in a setting where more expensive and labor intensive techniques are not feasible.The study will examine the safety and efficacy of two drug combinations (intrathecal morphine+fentanyl vs intrathecal morphine+bupivacaine) through a randomized control trial.

The investigators hypothesize that a single shot of either intrathecal morphine plus fentanyl or intrathecal morphine plus bupivacaine achieve analgesia and are safe in parturients experiencing normal labour.

ELIGIBILITY:
Inclusion Criteria:

* Parturients with singleton pregnancy
* Emancipated minors

Exclusion Criteria:

* Those who declined.
* Parturients with any identified complication of labour like preeclampsia, severe cardiac disease or previous operative delivery.
* Sepsis or wound at site of spinal injection.
* Allergy to any of the study drugs elicited from history.

Ages: 14 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia | 10 hours
  Monitoring the level of pain by the visual analogue scale to determine the total duration of analgesia in hours starting 5 min after drug administration

SECONDARY OUTCOMES:
APGAR score | 6 minutes
  The effect of the drugs to the fetus shall be determined by proxy from the APGAR scores of the baby determined at 1 minute and then at 5 minutes. Poor APGAR scores are those equal or less than seven (7).
Maternal side effects (composite) | 34 hours
  Maternal side effects including pruritis, urinary retention, high Bromage score, nausea and vomiting, abnormal blood pressure and pulse rate will be ascertained 24 hours after delivery.

OTHER OUTCOMES:
Degree of satisfaction | 24 hours after delivery
  Mothers would be asked if they were satisfied with their pain control during labor and if they would recommend to others
Time of onset of analgesia | After drug administartion
  Parturients would be monitored for when relief from pain was first felt.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kintu, M.med, Study Director — Department of Anesthesia and Critical Care, Makerere University, College of Health Sciences, Kampala,Uganda; Timothy Muyimbo, M.med, Principal Investigator — Department of Anesthesia and Critical Care, Makerere University, College of Health Sciences, Kampala,Uganda; Fred Bulamba, M.med, Study Chair — Department of Anesthesia and Critical Care, Makerere University, College of Health Sciences, Kampala,Uganda

REFERENCES:
- [Result] Decosterd I, Beggah AT, Durrer A, Buchser E. [Spinal opioids: mechanisms of action and chronic pain management]. Rev Med Suisse. 2006 Jun 21;2(71):1636-8, 1640. French. PMID 16878530
- [Result] Cascio M, Pygon B, Bernett C, Ramanathan S. Labour analgesia with intrathecal fentanyl decreases maternal stress. Can J Anaesth. 1997 Jun;44(6):605-9. doi: 10.1007/BF03015443. PMID 9187779
- [Result] Fontaine P, Adam P, Svendsen KH. Should intrathecal narcotics be used as a sole labor analgesic? A prospective comparison of spinal opioids and epidural bupivacaine. J Fam Pract. 2002 Jul;51(7):630-5. PMID 12160502